CLINICAL TRIAL: NCT05651854
Title: Effect of Bhramari Versus Sheetali Pranayama on Quality of Life in Hypertensive Patients
Brief Title: Effect of Different Pranayama Breathing Techniques on Quality of Life in Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Elsayed Mohammed Elsheikh, 7 ahmed elzayyat st, Dokki, Giza, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pranayama on hypertension
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-12

CONDITIONS: Hypertension; Stress; Aging Problems
Keywords: pranayama; quality of life; blood pressure; physical activity
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients are assigned randomly in groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bhramari pranayama breathing (Experimental): Bhrāmarī Prāṇāyāma breathing involves inhalation through both nostrils and producing humming sound of a bee while exhaling (Nivethitha et al., 2016).
  Interventions: Other: pranayama breathing
- Sheetali pranayama breathing (Experimental): Sheetali pranayama involve inhalation through extension of the tongue outside the mouth and roll the sides of the tongue up so that it would form a tube. At the end of inhalation, the tongue is drawn in, mouth is closed and exhale through the nose (Thanalakshmi et al., 2014).
  Interventions: Other: pranayama breathing

INTERVENTIONS:
Other: pranayama breathing — Bhramari and sheetali pranayama breathing

SUMMARY:
The purpose of the current study is to compare between the effect of Bhramari pranayama versus Sheetali pranayama on quality of life in hypertensive patients.

DETAILED DESCRIPTION:
People with hypertension have poorer sleep quality, less physical activity and more psychological stress than those with normal blood pressure. It has been shown that sleep affects vitality and health status and that sleep problems affect daily functioning and QOL, and so it can be assumed that in patients with hypertension, sleep problems will have a negative effect on QOL (Uchmanowicz et al., 2019).

Yogic breathing exercises are known as Pranayamas and are considered a form of meditation in itself, as well as a preparation for deep meditation. They promote physical well-being and self-awareness, improve lung and cognitive capacities, reduce blood pressure, anxiety, and other psychosomatic patterns, probably by increasing the parasympathetic tone. Pranayama alone has demonstrated numerous beneficial health effects, including stress relief, beneficial cardiovascular effect, improved respiratory function, and enhanced cognition (Jayawardena et al.,2020 ).

Since there is no study examined effect of Bhramari versus Sheetali on quality of life, physical fitness and stress in hypertensive elderly, this study aimed to examine this comparison.

ELIGIBILITY:
Inclusion Criteria:

- Sixty elderly are selected from both sexes. 2-Their age ranges from 60-75 years old. 3-Hypertensive patients (SBP is 140 -159 mmHg and/or DBP is 90-99 mmHg).

4-Their body mass index (BMI) ranged from < 30kg/m2. 5-All patients are medically stable.

Exclusion Criteria:

* - patients with cardiac problems e.g. atrial fibrillation, left bundle-branch block, heart failure, Recent myocardial infarction, coronary artery disease, or participation in cardiac rehabilitation following bypass surgery.

  2- Patients with history, symptoms of, and/or laboratory reports suggestive of renal, neurologic, or hepatic complications.

  3-Patients who have difficulty in rolling the tongue for Sheetali practice as stroke or Bell's palsy.

  4- Tongue swelling in case of acromegaly, amyloidosis, Myxedema and tongue cancer.

  5- Tongue pain in case of diabetic neuropathy, mouth ulcers, oral cancer and burn in the mouth.

  6- Chronic smokers and alcoholics. 7- Severe ear infections that interfere with bhramari breathing.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
cortisol | 3 months
  serum cortisol level

SECONDARY OUTCOMES:
Nitric oxide | 3 months
  serum nitric oxide
systolic blood pressure | 3 months
  systolic blood pressure
diastolic blood pressure | 3 months
  diastolic blood pressure
30 seconds sit to stand test | 3 months
  physical fitness assessment
SF12 quality of life questionnaire | 3 months
  quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Elnahas, professor doctor, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt